CLINICAL TRIAL: NCT01345747
Title: The Laryngeal Tube Suction vs Endotracheal Tube for Ventilation in Gynecological Laparoscopic Surgery
Brief Title: The Laryngeal Tube Suction Versus Endotracheal Tube for Ventilation in Gynecological Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Assistant Professor Nalinee Kovitwanawong, Department of Anesthesiology Faculty of Medicine Prince of Songkla University Thailand
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: LT-Laparo
Record Dates: First submitted 2011-04-25; First posted 2011-05-02 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Focus Groups
Keywords: laryngeal tube suction; gynecology; laparoscopic surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laryngeal tube (Experimental): laryngeal tube suction has suction port
  Interventions: Device: laryngeal tube (VBM Medizintechnik, Sulz, Germany)
- endotracheal tube (Experimental)
  Interventions: Device: laryngeal tube (VBM Medizintechnik, Sulz, Germany)

INTERVENTIONS:
Device: laryngeal tube (VBM Medizintechnik, Sulz, Germany) — laryngeal tube suction number 3 and 4
  Other Names: The laryngeal tube(VBM Medizintechnik, Sulz, Germany)

SUMMARY:
This study the investigators compare peak airway pressure (PAP), expire tidal volume (TV), end tidal CO2 (ETCO2), SpO2, mean arterial pressure (MAP) and heart rate (HR) after the insertion of laryngeal tube suction or endotracheal tube in patients undergoing elective gynecological laparoscopic surgery.

DETAILED DESCRIPTION:
Background:

For standard procedure, the endotracheal tube is used to ventilate the anesthetized patients who undergo gynecological laparoscopic surgery that increase intrabdominal pressure. Now there is a new supraglottic airway device, laryngeal tube suction (LTs) can be use instead of ETT.

Objective This study the investigators compare peak airway pressure (PAP), expire tidal volume (TV), end tidal CO2 (ETCO2), SpO2, mean arterial pressure (MAP) and heart rate (HR) after the insertion of laryngeal tube suction or endotracheal tube in patients undergoing elective gynecological laparoscopic surgery.

Material and methods Prospective single blinded randomized control trial, the patients were divided into two groups, LTs group and ETT group n = 60 for each group. All patients were induced anesthesia with fentanyl 1-2 mcg/kg, propofol 2 mg/kg, vecuronium 0.1 mg/kg then maintained anesthesia with air : oxygen 30%. Respirator setting are tidal volume 10 ml/kg, I/E 1:2 adjust RR base on ETCO2 keep ETCO2 35-40 mmHg.

Results No statistical difference in demographic data between groups. PAP and ETCO2 in the LTs group were significant higher than ETT group in the first 5 and 10 minutes but no statistically significant after 10 minutes until the end of operation. No statistically significant in TV and SpO2 between groups. In ETT group MAP and HR after insertion are significant higher than LTs group, no statistically significant about postoperative complication such as sorethroat, hoarseness and nausea vomiting.

Conclusion LTs can be used in gynecological laparoscopic surgery like ETT.

ELIGIBILITY:
Inclusion Criteria:

* female age between 20-65 years
* ASA class 1-2
* elective gynecologic laparoscopic surgery
* height < 180 cm
* BMI < 35 kg/m2

Exclusion Criteria:

* interincisor gap < 2.5 cm
* risk of aspiration
* history of difficult intubation
* oropharyngeal pathology
* allergy to anesthetic drug

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
respiratory parameter | 1-3 hours
  ETCO2, peak airway pressure and expired TV during operative period

SECONDARY OUTCOMES:
hemodynamic response | 30 minutes
  blood pressure and heart rate after LT insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand